CLINICAL TRIAL: NCT00573417
Title: A Placebo-Controlled Trial of Modafinil (Provigil) Added to Clozapine in Patients With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: North Suffolk Mental Health Association (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Donald Goff, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 34-02; Cephalon 670 Study
Record Dates: First submitted 2007-12-13; First posted 2007-12-14 (Estimated); Last update posted 2009-08-12 (Estimated); Status verified 2009-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Clozapine; Cognition; Metabolic Syndrome; Negative Symptoms; Wakefulness; Fatigue
MeSH Terms: conditions — Schizophrenia; Metabolic Syndrome; Fatigue | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- modafinil (Experimental): modafinil 100mg, 200mg, or 300mg (dose escalation)
  Interventions: Drug: modafinil
- placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: modafinil — modafinil 100mg tablets. dose excalation up to 300mg
  Other Names: Provigil
  Arms: modafinil
Drug: Placebo
  Arms: placebo

SUMMARY:
This pilot study is an eight-week, randomized, double-blind, placebo-controlled, escalating dose trial of the novel vigilance-promoting drug, modafinil, added to a stable dose of clozapine in 40 patients with schizophrenia or schizoaffective disorder. Modafinil will be initiated at 100 mg/d. After 2 weeks, the study drug may be increased to 200 mg/d and after 4 weeks, study drug may be increased to a maximum of 300 mg/d. Dose escalation will be based upon persistence of sedation versus emergence of side effects.

DETAILED DESCRIPTION:
This pilot study is an eight-week, randomized, double-blind, placebo-controlled, escalating dose trial of the novel vigilance-promoting drug, modafinil, added to a stable dose of clozapine in 40 patients with schizophrenia or schizoaffective disorder. Modafinil will be initiated at 100 mg/d. After 2 weeks, the study drug may be increased to 200 mg/d and after 4 weeks, study drug may be increased to a maximum of 300 mg/d. Dose escalation will be based upon persistence of sedation versus emergence of side effects.

1. Evaluate tolerability and safety of modafinil compared to placebo using the SAFTEE and vital signs.
2. Evaluate the effect size of modafinil compared to placebo upon wakefulness and fatigue using the Epworth Sleepiness Scale (ESS) and the Fatigue Severity Scale (FSS).
3. Evaluate the effect size of modafinil compared to placebo upon negative symptoms using the SANS total score.
4. Evaluate the effect size of modafinil compared to placebo upon cognitive functioning using a standard battery of cognitive tests.
5. Evaluate the effect size of modafinil compared to placebo upon weight, BMI, waist/hip circumference and fasting glucose and lipids.
6. Effect the variability of response in placebo and modafinil groups for each of the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Schizophrenia, any subtype or schizoaffective disorder
* Ages 18-65 years
* Capable of providing informed consent, or capable of providing assent with a guardian who provides informed consent
* Stable dose of clozapine for at least 1 month
* Three months of stable psychotic symptoms

Exclusion Criteria:

* Serious medical or neurological illness (unstable cardiac disease, seizure disorder, malignancy, liver or renal impairment, etc.)
* Current substance abuse
* Pregnancy, nursing, or unwilling to use appropriate birth control measures during participation if female and fertile.
* Unable to complete neuropsychological tests
* History of serious blood dyscrasia requiring discontinuation of clozapine
* Serious suicidal or homicidal risk within the past six months
* Current treatment with a psychostimulant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-09; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect size of modafinil compared to placebo upon cognitive functioning using a standard battery of cognitive tests. | 8 weeks

SECONDARY OUTCOMES:
Evaluate tolerability and safety of modafinil compared to placebo using the SAFTEE and vital signs. | 8 weeks
Evaluate the effect size of modafinil compared to placebo upon wakefulness and fatigue using the Epworth Sleepiness Scale (ESS) and the Fatigue Severity Scale (FSS). | 8 weeks
Evaluate the effect size of modafinil compared to placebo upon negative symptoms using the SANS total score. | 8 Weeks
Evaluate the effect size of modafinil compared to placebo upon weight, BMI, waist/hip circumference and fasting glucose and lipids. | 8 weeks
Effect the variability of response in placebo and modafinil groups for each of the outcome measures. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Donald Goff, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Freedom Trail Clinic, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Freudenreich O, Henderson DC, Macklin EA, Evins AE, Fan X, Cather C, Walsh JP, Goff DC. Modafinil for clozapine-treated schizophrenia patients: a double-blind, placebo-controlled pilot trial. J Clin Psychiatry. 2009 Dec;70(12):1674-80. doi: 10.4088/JCP.08m04683. Epub 2009 Aug 11. PMID 19689921